CLINICAL TRIAL: NCT05325996
Title: Evaluating Effectiveness of Home Testing Devises for Assisting in Management of Glaucoma Outside a Clinical Setting During a 2 Year Period.
Brief Title: Evaluating Home Testing Devices for the Management of Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, M. Reza Razeghinejad MD, Principal Investigator, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB# 2021-79
Record Dates: First submitted 2022-03-25; First posted 2022-04-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma, Open-Angle
Keywords: Open Angle Glaucoma; Perimetery; Tonometry; Eye Pressure; Visual Field; Home Test
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Moderate Glaucoma (Experimental): Subjects between ages 20-80 years with a diagnosis of mild and moderate Open Angle Glaucoma in at least one eye with 20/50 vision or better will be included in this study. All subjects will have the Olleyes Perimeter measure their own visual acuity and field once a week during a 2 year period and iCare home to measure their eye pressure 3 times a day for 7 days every 3 months during a 2 year period.
  All patient will have their routine glaucoma assessment with the standard 24-2 Automatic Perimetry Humphrey Field Analyzer at baseline and every 6 months during a 2 year period; and Spectralis Optical Coherence Tomography thickness of peripapillary RNFL and macular ganglion cell at baseline and yearly during a 2 year period.
  Interventions: Diagnostic Test: Standard Automatic Perimetry Humphrey Field Analyzer; Diagnostic Test: visuALL H; Diagnostic Test: iCare Home Tonometer; Diagnostic Test: Spectralis Optical coherence tomography (OCT)

INTERVENTIONS:
Diagnostic Test: Standard Automatic Perimetry Humphrey Field Analyzer — Standard Automatic Perimetry (SAP) using the Swedish Interactive Threshold Algorithm (SITA) Standard Strategy measures the visual field in an ophthalmic setting.
  Other Names: SAP HFA
Diagnostic Test: visuALL H — visuALL H a new portable perimeter measuring the visual field and acuity in a non ophthalmic setting.
Diagnostic Test: iCare Home Tonometer — iCare HOME tonometer is a device developed for patients/subjects to measure their eye pressure at home.
Diagnostic Test: Spectralis Optical coherence tomography (OCT) — Optical coherence tomography (OCT) is a computerized picture measuring the thickness of the inner layer of the retina that makes the optic nerve.

SUMMARY:
With the advancement in technology we have the opportunity of performing the glaucoma testing at home to monitor the disease. The purpose of this study is evaluating the feasibility and patient acceptance of home testing with head mounted perimetry; detection of progression with head mounted perimetry vs office based perimetry; and monitoring the eye pressure measured by patients at home using a portable tonometer.

DETAILED DESCRIPTION:
Standard Automatic Perimetry (SAP) is the gold standard test for evaluation of diseases of the visual pathway like glaucoma. Its main goal is to measure differential light sensitivity at several locations in the field of vision. Several devices have been developed since the advent of the Octopus Perimeter and the Humphrey Field Analyzer (HFA) is now the most commonly used machine for checking the visual field. These devices have a number of disadvantages including being stressful for debilitated, ill, or elderly patients to keep their heads still in the perimeter bowl during the test.

Recently, several methods have been introduced for checking the visual field using laptops or iPads. These modalities bring portability but lack fixation methods, environmental control, hardware standardization, and lack the ability of checking the visual acuity. These deficiencies may limit their wide usage. VisuALL is a Head Mounted perimeter that connects to its application on the cell phone or tablet via Bluetooth. In addition to being a portable perimeter and checking visual acuity, it has the ability of monitoring fixation with an accuracy of 1 degree. The measured visual field will be saved on a cloud space and available to the physician and patient. It has been shown that the more frequent visual tests we perform, the earlier we would be able to detect visual field progression. Currently, the visual field test is performed on patients in an ophthalmology clinic with a technician present during the test. The VisuALL has a demo video to provide education to the patient on the simple and user-friendly process of visual field testing.

Tonometry is the measurement of eye pressure. iCare Home Tonometer measurements have been shown to be highly correlated to Goldmann Tonometer measurements which are performed in the ophthalmic office. Multiple studies have highlighted the shortcomings of relatively infrequent in office tonometry. Recent studies have suggested that peak out of office eye pressures are often higher than in office pressures and the iCare Home Tonometer is one option to assess eye pressure outside of the office.

Home monitoring of glaucoma may present opportunities to reduce the burdens of office visits while increasing the monitoring of the visual field and eye pressure. This study is intended to assess the feasibility and utility of home based perimetry and tonometry in the management of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80 years
2. Mild and Moderate Open Angle Glaucoma (OAG)
3. Refraction under 12.00 diopter of spherical refractive error and astigmatism of less than 2.5 diopter.

Exclusion Criteria:

1. Spherical refraction outside > ± 12.00 D and cylinder correction > +2.5 D.
2. Visual acuity worse than 20/50 either eye
3. Cataract surgery with or without Minimally Invasive Glaucoma Surgery (MIGS) less than 90 days prior to enrollment
4. Filtering surgeries less than 6 months prior to enrollment
5. Intraocular surgery other than:

   1. Non-complicated MIGS more than 90 days prior to enrollment;
   2. Cataract or refractive surgery performed more than 90 days before enrollment and without posterior capsule opacification
   3. Other glaucoma surgery more than 6 months prior to enrollment.
6. History of systemic or ocular condition (other than glaucoma or mild to moderate cataract) known to affect visual function.
7. History of medication known to affect visual function or influence patient reaction time
8. Inability to use device after remote training session
9. Subjects unwilling and/or unable to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Visual Field Mean Deviation with VisuALL | 12 minutes each week for 104 weeks
  The visual field measures sensitivity of the retina to light at several locations in the peripheral vision. The difference of mean of these measurements compared to a normal database is presented in negative or positive values called mean deviation.
  Visual field mean deviation (MD) (light measurement in decibels in multiple spots across the central and peripheral retina known as entire visual field) will be captured by VisuALL per eye once a week during a 2 year period at participant's home.
Change in Intraocular Pressure with iCare | 15 minutes daily over 1 week, 8 times for 2 years
  Intraocular pressure, measured in millimeters of mercury (mmHG), will be measured by patients using a device called iCare Home Tonometer, specifically designed for patients to measure their eye pressures at home. They will measure eye pressure of each eye 3 times a day for 7 days every 3 months during a 2 year period at participant's home.

SECONDARY OUTCOMES:
Change in Visual Field Mean Deviation with Humphrey Field Analyzer | 2 hours, 5 times for 2 years
  The visual field measures sensitivity of the retina to light at several locations in the peripheral vision. The difference of mean of these measurements compared to a normal database is presented in negative or positive values called mean deviation.
  Visual field mean deviation (MD) (light measurement in decibels in multiple spots across the central and peripheral retina known as entire visual field) will be measured in the office by Humphrey perimeter 24-2 SITA standard per 3 times at baseline and then every 6 months during a 2 year period..

OTHER OUTCOMES:
Change in Retinal Nerve Fiber Layer (RNFL) Thickness | 10 minutes, 3 times for 2 years
  Retinal Nerve Fiber Layer (RNFL) Thickness in microns will be obtained by a computerized picture without touching the eye with Spectralis (Zeiss) Optical Coherence Tomography (OCT) at baseline and then yearly during a 2 year period.

CONTACTS AND LOCATIONS:
Overall Officials: M. Reza Razeghinejad, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No